CLINICAL TRIAL: NCT00559936
Title: Effectiveness and Safety of Topical Bevacizumab (Avastin) for Treatment of Corneal Neovascularization
Brief Title: Topical Avastin for Treatment of Corneal Neovascularization
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Principal Investigator, Reza Dana, MD, Director, Cornea and Refractive Surgery Service, Massachusetts Eye and Ear Infirmary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-12-077; 06-12-077 (Other: Massachusetts Eye and Ear Infirmary)
Record Dates: First submitted 2007-11-14; First posted 2007-11-16 (Estimated); Results first posted 2012-09-24 (Estimated); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Corneal Neovascularization
MeSH Terms: conditions — Corneal Neovascularization | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Topical Avastin 1.0% (Experimental): Each patient will receive topical Avastin in one eye.
  Interventions: Drug: Topical Avastin 1%

INTERVENTIONS:
Drug: Topical Avastin 1% — Avastin (bevacizumab) 1%
  Other Names: bevacizumab

SUMMARY:
The purpose of this study is to determine the effectiveness and safety of Topical Bevacizumab (Avastin) for treatment of corneal neovascularization.

DETAILED DESCRIPTION:
Primary outcomes measures included neovascular area (NA), defined as the area of the corneal vessels themselves; vessel caliber (VC), defined as the mean diameter of the corneal vessels; and invasion area (IA), defined as the fraction of the total cornea into which the vessels extend. The occurrence of ocular and systemic adverse events was closely monitored throughout the course of the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, at least 18 years of age
* Clinical stable corneal neovascularization (as defined above)
* Ability to understand and provide informed consent to participate in this study and willingness to follow study instructions and likely to complete all required visits.
* All female patients of childbearing potential will be excluded. A female is considered to be of childbearing potential unless she is postmenopausal and without menses for 12 months or without a uterus and/or both ovaries.

Exclusion Criteria:

* Current or recent (≤ 1 month) systemic corticosteroid therapy or periocular corticosteroid injections to the study eye
* Current or recent (≤ 3 months) intravitreal drug injection to the study eye; recent (≤ 1 month) change in dose and frequency of topical steroids and/or non-steroidal anti-inflammatory agents
* Uncontrolled hypertension defined as systolic blood pressure of ≥ 150 mmHg or diastolic blood pressure of ≥ 90 mmHg; history of a thromboembolic event, including myocardial infarction or cerebral vascular accident
* Patients age 75 or older; history of renal abnormalities
* Recent (≤ 3 months ) or planned surgery
* History of coagulation abnormalities, including end stage liver disease or current anticoagulation medication other than aspirin (warfarin, heparin, enoxaparin, or similar anticoagulant agent)
* All female patients of childbearing potential (a female is considered to be of childbearing potential unless she is postmenopausal and without menses for 12 months or without a uterus and/or both ovaries)
* Any condition (including language barrier) that precludes patient's ability to comply with study requirements including completion of study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-02; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Reza Dana, M.D., MPH, Principal Investigator — Massachusetts Eye and Ear Infirmary
Locations (1):
- Massachusetts Eye and Ear Infirmary, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Cheng SF, Dastjerdi MH, Ferrari G, Okanobo A, Bower KS, Ryan DS, Amparo F, Stevenson W, Hamrah P, Nallasamy N, Dana R. Short-term topical bevacizumab in the treatment of stable corneal neovascularization. Am J Ophthalmol. 2012 Dec;154(6):940-948.e1. doi: 10.1016/j.ajo.2012.06.007. Epub 2012 Sep 8. PMID 22967868
- [Derived] Dastjerdi MH, Al-Arfaj KM, Nallasamy N, Hamrah P, Jurkunas UV, Pineda R 2nd, Pavan-Langston D, Dana R. Topical bevacizumab in the treatment of corneal neovascularization: results of a prospective, open-label, noncomparative study. Arch Ophthalmol. 2009 Apr;127(4):381-9. doi: 10.1001/archophthalmol.2009.18. PMID 19365012

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Cornea Service at Massachusetts Eye and Ear Infirmary from February 2007 through October 2010.
Pre-assignment Details: Only patients with superficial or deep corneal neovascularization that extends farther than 2 mm from the limbus will be considered.
Period: Overall Study
Arm/Group | Topical Avastin 1.0%
Started | 24
Completed | 20
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Topical Avastin 1.0%
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.5 (3.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 16
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: The Size and Extent of Corneal Neovascularization Will be Measured by Computerized Image Analysis of Corneal Photographs Taken Throughout the Study.
Description: The efficacy of bevacizumab in the treatment of corneal NV was evaluated by comparing corneal photographs taken at baseline with corneal photographs taken at the follow-up visits. Percent change from baseline was measured.
Time Frame: Six Months
Population: Participants who received investigational treatment were analyzed.
Measure: Mean (Standard Deviation); unit: percent change since baseline
Arm/Group | Topical Avastin 1.0%
Number analyzed (Participants) | 20
percent change since baseline | 27.9 (9.2)

2. Primary Outcome: Ocular and Systemic Safety
Description: The occurrence of ocular and systemic adverse events was closely monitored over the course of this study. Ocular adverse events were monitored through complete ocular examinations including visual acuity measurement, intraocular pressure measurement, biomicroscopy, and corneal fluorescein staining. Systemic adverse events were identified with physical examinations, patient questioning, and blood pressure measurements taken throughout the study period.
Time Frame: All study visits
Population: Participants treated with investigational medication were analyzed.
Measure: Number; unit: participants
Arm/Group | Topical Avastin 1.0%
Number analyzed (Participants) | 20
participants | 0

ADVERSE EVENTS:
Arm/Group | Topical Avastin 1.0%
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes